CLINICAL TRIAL: NCT01213199
Title: Efficacy and Safety of Adapalene Gel 0.3% in the Treatment of Atrophic Acne Scars. A Pilot Study.
Brief Title: Adapalene Gel 0.3% in the Treatment of Atrophic Acne Scars
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.03.SPR.29088
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2015-03

CONDITIONS: Acne Scars
MeSH Terms: interventions — Adapalene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Differin 0.3% (Experimental): Differin® 0.3% Gel
  Adapalene 0.3%
  Topical to the face, once daily application in the evening for the first four weeks and twice daily application in the morning and in the evening for the following 20 weeks.
  Interventions: Drug: Adapalene

INTERVENTIONS:
Drug: Adapalene — Adapalene Gel 0.3%
  Other Names: Differin 0.3%

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Adapalene Gel 0.3% in the treatment of atrophic acne scars.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any race, aged 18 to 50 years inclusive
* Subjects with a past history of acne and with moderate to severe facial atrophic acne scars

Exclusion Criteria:

* Subjects with active inflammatory acne lesions
* Subjects with hypertrophic acne scars

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha J. Patel, MD, Principal Investigator — Johns Hopkins Medical Institut
Locations (1):
- Manisha PATEL, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Loss MJ, Leung S, Chien A, Kerrouche N, Fischer AH, Kang S. Adapalene 0.3% Gel Shows Efficacy for the Treatment of Atrophic Acne Scars. Dermatol Ther (Heidelb). 2018 Jun;8(2):245-257. doi: 10.1007/s13555-018-0231-8. Epub 2018 Mar 16. PMID 29549598
- See also: Related Info — http://galderma.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in =25 March 2011, last patient out= 21 Sep 2012
Groups:
- Differin® 0.3% Gel: Differin® 0.3% Gel Adapalene 0.3%
  Topical to the face Once daily application in the evening for the first 4 weeks and twice daily application in the morning and in the evening for the following 20 weeks.
Period: Overall Study
Arm/Group | Differin® 0.3% Gel
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Analysis population includes all 20 subjects enrolled into the study (Intent-to-Treat population).
Arm/Group | Differin® 0.3% Gel
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Global Scarring Severity
Description: Grade Level:
  1. Macular disease
  2. Mild disease
  3. Moderate disease
  4. Severe disease
Time Frame: Week 24
Population: The analysis population includes 18 subjects whose data were available at this time frame (week 24).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Differin® 0.3% Gel
Number analyzed (Participants) | 18
units on a scale | 2.7 (0.8)

ADVERSE EVENTS:
Arm/Group | Differin® 0.3% Gel
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No